CLINICAL TRIAL: NCT05052333
Title: An International Study Examining the Psychosocial Impacts of COVID-19 Pandemic.
Brief Title: Examine the Psychosocial Impacts of COVID-19 Pandemic.
Status: Completed | Type: Observational
Sponsor: University of Otago (Other)
Collaborators: International Islamic University, Islamabad (Other); Universitas Ahmad Dahlan (Other); Gadjah Mada University (Other); Ibn Sina University of Medical and Pharmaceutical Sciences, Iraq (Other); Al-Mustansiriyah University (Other); Hasan Kalyoncu University (Other); University of Washington (Other); University of Malaya (Other); University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Sandila Tanveer, Assistant Research Fellow, University of Otago
Other Study IDs: UOtago
Record Dates: First submitted 2021-09-19; First posted 2021-09-22 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Psychosocial Impacts; COVID-19 Pandemic
Keywords: Psychological distress; Wellbeing; Mental health; Reliability and validity; Low and middle income countries; Cross-cultural comparisons
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Examining the psychosocial impacts of COVID-19 in Pakistan.: This is exploratory research and data will be obtained on a set of measures using a bilingual (Urdu-English) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of COVID-19 in Iraq.: This is exploratory research and data will be obtained on a set of measures using a bilingual (Arabic-English) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of COVID-19 in Türkiye.: This is exploratory research and data will be obtained on a set of measures using a unilingual (Turkish) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of COVID-19 in Iran.: This is exploratory research and data will be obtained on a set of measures using a Bilingual (Persian-English) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of COVID-19 in Malaysia.: This is exploratory research and data will be obtained on a set of measures using a bilingual (Malay-English) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of COVID-19 in Indonesia.: This is exploratory research and data will be obtained on a set of measures using a unilingual (Indonesian) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.
- Examining the psychosocial impacts of Covid-19 in Somaliland.: This is exploratory research and data will be obtained on a set of measures using a unilingual (Somalia) survey. No predefined conditions apply to explain the nature of the study group other than inclusion and exclusion criteria.

SUMMARY:
This is an observational study examining the psychosocial impacts of the COVID-19 pandemic in seven low-and-middle income countries (Indonesia, Iran, Iraq, Malaysia, Pakistan, Somaliland, and Turkiye). The data was obtained on standardised measures of wellbeing (WHO Well-Being Index), psychological distress (Kessler 10), post-traumatic stress (PTSD Checklist for DSM-5), post-traumatic growth (Posttraumatic Growth Inventory), and a novel pandemic-related stress (COVID Psychosocial Impacts Scale). Data was collected employing either a unilingual (in native language) or bilingual online survey (with English as a second language) from participants (N=2574) aged 18 and above using a non-probability convenient sampling. The findings enabled us to examine the psychosocial impacts of COVID-19, validate the translations of the CPIS and standardized measures; and determine the trajectory of study variables with pandemic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Currently residing in the country of interest.
* Additional inclusion criterion applies to bilingual studies; which is having English as a second language.

Exclusion Criteria:

* Aged below 18 years.
* Not residing in the country of interest.
* Additional exclusion criterion applies to bilingual studies; which is not having English as a second language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the general population using convenience sampling in each of the seven locations (Indonesia, Iran, Iraq, Malaysia, Pakistan, Somaliland, and Turkiye). The specific details (e.g., residents of a certain town) may vary from country to country and it will be outlined by the international collaborators in local ethics applications.
Sampling Method: Non-Probability Sample
Enrollment: 2574 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Examining the psychosocial impacts of the COVID-19 pandemic. | Data was collected in a short-time window on each site. The time of data collection varies across site and was collected from Dec 2021 to Sep 2023.
  To explore the psychosocial impacts of the COVID-19 pandemic on self-report measures of wellbeing (WHO-5), psychological distress (K10), post-traumatic stress (PCL-5), post-traumatic growth (PTGI), and pandemic-related stress (CPIS) in seven LMICs. The data will be collected employing a unilingual (Indonesia, Somaliland, Turkey) or bilingual (Iran, Iraq, Malaysia, Pakistan) survey. With-in-subjects and between-subjects designs together with exploratory regression analyses will be employed to characterize this outcome.

OTHER OUTCOMES:
Analyzing the psychometric properties of the translations of the newly developed CPIS and other standardized measures. | The time of data collection varies across site and was collected from Dec 2021 to Sep 2023.
  The findings will give psychometric information on the translations and suitability of use of the newly developed CPIS and other standardized questionnaires (K10, WHO-5, PCL-5, PTGI) in seven LMICs. The metric used to characterize this outcome involves reliability (internal consistency) and validity (construct) analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Bell, MD, Principal Investigator — University of Otago Christchurch, New Zealand; Sandila Tanveer, PhD, Principal Investigator — University of Otago Christchurch, New Zealand; Ruqayya Sulaiman-Hill, PhD, Principal Investigator — University of Otago Christchurch, New Zealand; Richard Porter, MRCPsych, Study Director — University of Otago Christchurch, New Zealand; Joseph Boden, PhD, Principal Investigator — University of Otago Christchurch, New Zealand; Ben Beaglehole, FRANZCP, Principal Investigator — University of Otago Christchurch, New Zealand; Shaystah Dean, PhD, Principal Investigator — University of Otago Wellington, New Zealand; Philip Schluter, PhD, Principal Investigator — University of Canterbury, New Zealand
Locations (9):
- University of Washington, Seattle, Washington, United States
- Indonesia (2):
  - Universitas Ahmad Dahlan, Yogyakarta
  - Universitas Gadjah Mada, Yogyakarta
- University of Social Welfare and Rehabilitation Sciences, Tehran, Iran
- Iraq (2):
  - Ibn Sina University of Medical and Pharmaceutical Sciences, Baghdad
  - Mustansiriyah University, Baghdad
- Universiti Malaya, Kuala Lumpur, Malaysia
- International Islamic University, Islamabad, Pakistan
- Hasan Kalyoncu Üniversitesi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bell C, Beaglehole B, Bell R, Tanveer S, Sulaiman-Hill R, Boden J, Porter R. Learning from previous disasters: Potential pitfalls of epidemiological psychosocial research in the COVID-19 environment. Aust N Z J Psychiatry. 2021 Jul;55(7):646-649. doi: 10.1177/0004867421998783. Epub 2021 Mar 1. PMID 33645256
- [Background] Bell C, Williman J, Beaglehole B, Stanley J, Jenkins M, Gendall P, Rapsey C, Every-Palmer S. Challenges facing essential workers: a cross-sectional survey of the subjective mental health and well-being of New Zealand healthcare and 'other' essential workers during the COVID-19 lockdown. BMJ Open. 2021 Jul 19;11(7):e048107. doi: 10.1136/bmjopen-2020-048107. PMID 34281926
- [Background] Fergusson DM, Boden JM, Horwood LJ, Mulder RT. Perceptions of distress and positive consequences following exposure to a major disaster amongst a well-studied cohort. Aust N Z J Psychiatry. 2015 Apr;49(4):351-9. doi: 10.1177/0004867414560652. Epub 2014 Nov 27. PMID 25430912
- [Background] Jenkins M, Hoek J, Jenkin G, Gendall P, Stanley J, Beaglehole B, Bell C, Rapsey C, Every-Palmer S. Silver linings of the COVID-19 lockdown in New Zealand. PLoS One. 2021 Apr 1;16(4):e0249678. doi: 10.1371/journal.pone.0249678. eCollection 2021. PMID 33793672
- [Background] Kessler RC, Barker PR, Colpe LJ, Epstein JF, Gfroerer JC, Hiripi E, Howes MJ, Normand SL, Manderscheid RW, Walters EE, Zaslavsky AM. Screening for serious mental illness in the general population. Arch Gen Psychiatry. 2003 Feb;60(2):184-9. doi: 10.1001/archpsyc.60.2.184. PMID 12578436
- [Background] Tedeschi RG, Cann A, Taku K, Senol-Durak E, Calhoun LG. The Posttraumatic Growth Inventory: A Revision Integrating Existential and Spiritual Change. J Trauma Stress. 2017 Feb;30(1):11-18. doi: 10.1002/jts.22155. Epub 2017 Jan 18. PMID 28099764
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Tanveer S, Schluter PJ, Beaglehole B, Porter RJ, Boden J, Sulaiman-Hill R, Scarf D, Dean S, Assad F, Hasnat MA, Bell C. The COVID Psychosocial Impacts Scale: A Reliable and Valid Tool to Examine the Psychosocial Impacts of the COVID-19 Pandemic. Int J Environ Res Public Health. 2023 May 29;20(11):5990. doi: 10.3390/ijerph20115990. PMID 37297593
- [Result] Tanveer S, Schluter PJ, Porter RJ, Boden J, Beaglehole B, Sulaiman-Hill R, Dean S, Bell R, Al-Hussainni WN, Arshi M, Amer Nordin AS, Dinc M, Khan MJ, Khoshnami MS, Majid Al-Masoodi MA, Moghanibashi-Mansourieh A, Noruzi S, Rahajeng A, Shaikh S, Tanveer N, Topcu F, Yapan S, Yunianto I, Zoellner LA, Bell C. Examining the psychosocial impacts of the COVID-19 pandemic: an international cross-sectional study protocol. BMJ Open. 2023 Apr 12;13(4):e067886. doi: 10.1136/bmjopen-2022-067886. PMID 37045574
- See also: World Health Organization (2021). Mental Health and Psychosocial Considerations During the COVID-19 Outbreak. — https://apps.who.int/iris/handle/10665/331490
- See also: The Coronavirus Health Impact Survey (2019) — http://www.crisissurvey.org/